CLINICAL TRIAL: NCT06097182
Title: Post-biotic Intervention for Acute Stress Management
Acronym: PIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Jeroen Schmitt, Senior Principal Scientist, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-086
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stress Response; Mood State; Sleep; Cognition
Keywords: gut-brain-axis; stress response; Cognition; Mood State; Sleep
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Study design: The study will be carried out according to a randomized, placebo-controlled, double-blind, 3 arm parallel-groups design. It will be executed as a hybrid study (partially decentralized). Total study duration is 9 days (day 0 to day 8), excluding screening and enrolment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-biotic, colonic delivery (Experimental): n=25, 250mg post-biotic once daily in a polymer coated vegan gelatine capsule (colonic delivery)
  Interventions: Dietary Supplement: Post-biotic (Colonic-Delivery capsule); Other: Placebo
- Post-biotic, regular administration (Active Comparator): n=25, 250mg post-biotic once daily in a regular uncoated vegan gelatine capsule
  Interventions: Dietary Supplement: Post-biotic (Regular Administration capsule); Other: Placebo
- Placebo (Placebo Comparator): n=25, 250mg Maltodextrin once daily in a regular uncoated vegan gelatine capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Post-biotic (Colonic-Delivery capsule) — 250mg post-biotic once daily in a polymer coated vegan gelatine capsule (colonic delivery)
  Arms: Post-biotic, colonic delivery
Dietary Supplement: Post-biotic (Regular Administration capsule) — 250mg post-biotic once daily in a regular uncoated vegan gelatine capsule
  Arms: Post-biotic, regular administration
Other: Placebo — 250mg Maltodextrin once daily in a regular uncoated vegan gelatine capsule

SUMMARY:
The study aims to evaluate the sub-chronic effects of colonic delivery of a post-biotic on stress response, mood state, sleep, and cognition in healthy young subjects with elevated self-reported stress levels. It is hypothesized that oral intake of the post-biotic, when released in the colonic intestinal site, leads to a blunted subjective and objective stress response after a stress induction.

DETAILED DESCRIPTION:
Scientific findings over the past years suggest that certain bacteria in our gastrointestinal system have an influence on our mood, although, the mechanisms are not yet well understood. One of the possibilities is that bacteria produce compounds that interact with neurons in the gut. These neurons could subsequently send signals to the brain.

This study is a proof of principle study examining the effects of a post-biotic in the distal intestinal tract (terminal ileum, colon) on stress response, mood state, sleep, and cognition. The study is expected to provide key insights in the potential of treatment strategies aimed at stimulating the colonic enteric nervous system to exert mood enhancement. It is hypothesized that interactions with the local Enteric Nervous System leading to stress reduction, mood enhancement and sleep promotion effects. The study will employ an in-person clinic visit, in addition to traditional self-reported, behavioural, and physiological outcome measures; exploratory digital health outcomes will also be included to identify novel objective mood/stress measures.

This study seeks to recruit a total of 75 healthy males (25 in each arm), between the ages of 21-30 years old (inclusive) from local community outreach in Singapore over a period 12 months. This study is a hybrid study (partially decentralized).

The total duration of participation from each participant will be 9 days (excluding, the screening and enrolment days).

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 30 years
* Men
* Perceived Stress Scale (PSS-10) score >13
* Own and uses a smartphone that is capable to run the study applications with access to the internet
* Adequate fluency in the English language to understand the inform consent process, study instructions and study assessments
* Sufficient vision and hearing to complete study procedures
* Willing to commit to the study procedures
* Willing and able to participate and to give written informed consent All inclusion criteria will be assessed based on self-reported information during the screening visit.

Exclusion Criteria:

* Past (< 6 months prior to the study) or current major neurological, psychiatric, gastrointestinal, metabolic disease or cardiovascular disease
* Past (<1 months prior to the study) or current use of psychoactive medication, cardiovascular medication, or corticosteroids.
* Known medical history of hypotension or currently on antihypertensive medication
* Alcohol intake >1 units day
* Present or past history of alcohol or drug addiction and/or recreational drug use
* BMI <18.5 or >25 kg/m2
* Maltodextrin allergy
* Members of the research team or their immediate family members. An immediate family member is defined as spouse, parent, child, or sibling, whether biological or legally adopted All exclusion criteria will be assessed based on self-reported information during the screening call.

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol | Day 7 (5/day)
  cortisol levels, as a marker of hypothalamic-pituitary-adrenal (HPA) axis activation

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI-6) | Day 7 (2/day)
  The STAI-6 is a validated short-form version (6 items) of the 40-item STAI questionnaire, measuring current anxiety symptoms on a 4-point Likert scale. Total score is calculated (range 6-24).
The Brunel Mood Scale (BRUMS) | Day 7 (2/day)
  The BRUMS is a 24-item questionnaire of simple mood descriptors such as angry, nervous, unhappy, and energetic. The BRUMS has six subscales, with each of the subscales containing four mood descriptors. The subscales are anger, confusion, depression, fatigue, tension, and vigour. Responses are recorded using a 5-point Likert scale (0-4).
Heart Rate | Days 1-7
  Measured as beats per minute. Continuous monitoring via a smart-watch.
Sleep Activity | Days 1-7
  During sleep, the activity will be monitored via a smart-watch throughout the sleep session.

OTHER OUTCOMES:
Ecological Momentary Assessments (EMA) | Day 1-6 (4/day), Day 7 (2/day), Day 8 (1/day)
  Subjects are asked to indicate their current state on a visual analogue scale ranging from 'not at all' to 'very much' using a slider.
Salivary α-amylase | Day 7 (5/day)
  α-amylase levels, as a marker of autonomic nervous system activation
Gastrointestinal Symptoms | Days 1-7 (1/day)
  Participants will be asked to rate the average severity of the following five symptoms over the preceding 24 hours on a 5-point scale from 0 (absent) to 4 (very severe): bloating/distension, passage of gas, rumbling, feeling of fullness and abdominal discomfort/pain. A daily total score is calculated by summing all items recorded each day. A lower score is concomitant with lower severity of symptoms.
Respiratory Rate | Days 1-7
  Measured as how many breaths per minute. Continuous monitoring via a smart-watch.
Electrodermal Activity (EDA) | Days 1-7
  4 user-initiated 2 min sessions per day. Measured via a smart-watch and the total score per session is provided by the watch.
Speech Analysis for digital stress biomarkers | Day 7 (2/day)
  Subjects are requested to verbally reproduce an orally presented standard short story from Newcomer Story Set. A high-resolution video with audio will be recorded and exploratory analyses of speech characteristics will be performed.
Eye Movement Analysis for digital stress biomarkers | Day 7 (2/day)
  Subjects are requested to verbally reproduce an orally presented standard short story from Newcomer Story Set. A high-resolution video with audio will be recorded and exploratory analyses of eye movements will be performed.
Facial Expression Analysis for digital stress biomarkers | Day 7 (2/day)
  Subjects are requested to verbally reproduce an orally presented standard short story from the Newcomer Story Set. A high-resolution video with audio will be recorded and exploratory analyses of facial characteristics will be performed.
Handwriting Analysis for digital stress biomarkers | Day 7 (2/day)
  Subjects are requested to write down words of a specific category with a specified starting letter. As an exploratory outcome, a digital picture of the written text will be analyzed for handwriting characteristics such as trace, calibre, slant, and distance.
Cognitive performance | Days 1-8
  Cognitive performance will be assessed with a short (5 min) test battery consisting of tests of processing speed, spatial memory, and reaction time delivered through a mobile application that was developed to assess individuals' cognition in natural, non-laboratory, settings.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Schmitt, PhD, Principal Investigator — Singapore Institute of Clinical Sciences (SICS), A*STAR
Locations (1):
- Human Development Research Centre, SICS, A*STAR, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boets E, Gomand SV, Deroover L, Preston T, Vermeulen K, De Preter V, Hamer HM, Van den Mooter G, De Vuyst L, Courtin CM, Annaert P, Delcour JA, Verbeke KA. Systemic availability and metabolism of colonic-derived short-chain fatty acids in healthy subjects: a stable isotope study. J Physiol. 2017 Jan 15;595(2):541-555. doi: 10.1113/JP272613. Epub 2016 Sep 18. PMID 27510655